CLINICAL TRIAL: NCT06903988
Title: A Randomized Controlled Study on the Efficacy and Safety of Laparoscopic Lateral Suspension and Transvaginal Sacrospinous Ligament Fixation in Patients With Pelvic Organ Prolapse
Brief Title: Efficacy and Safety of Laparoscopic Lateral Suspension and Transvaginal Sacrospinous Ligament Fixation in Patients With Pelvic Organ Prolapse
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wang Shiyan, Associate Chief Physician, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024PHB374-002
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Organ Prolapse (POP)
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic lateral suspension (Experimental)
  Interventions: Procedure: laparoscopic lateral suspension
- transvaginal sacrospinous ligament fixation (Active Comparator)
  Interventions: Procedure: Transvaginal sacrospinous ligament fixation

INTERVENTIONS:
Procedure: laparoscopic lateral suspension — Laparoscopic lateral suspension: Place a 1/2 T4 mesh in the vesicovaginal space. The two lateral slings are passed out from the outer upper side of the bilateral anterior superior iliac spine, and the prolapsed organs are suspended to the abdominal wall.
  Arms: laparoscopic lateral suspension
Procedure: Transvaginal sacrospinous ligament fixation — Transvaginal sacrospinous ligament fixation: Dissect the rectovaginal space to expose the right sacrospinous ligament, and fix the cervix or vaginal cuff to the right sacrospinous ligament.
  Arms: transvaginal sacrospinous ligament fixation

SUMMARY:
This study is a single-center, non-blinded, non-inferiority randomized controlled trial, planning to recruit 86 patients with Stage III or higher pelvic organ prolapse who are unresponsive to conservative treatment and are requesting surgical treatment. Patients who meet the inclusion and exclusion criteria will be randomly assigned to the transvaginal sacrospinous ligament fixation group and the laparoscopic lateral suspension group in a 1:1 ratio. Follow-ups will be conducted at 1 month, 3 months, 6 months, and 1 year after surgery for the enrolled patients. The primary outcome measure is the difference in surgical success rate between the two groups of patients at 1 year after surgery. We hypothesize that the surgical success rate of laparoscopic lateral suspension is not inferior to that of transvaginal sacrospinous ligament fixation

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. According to the POP-Q classification, patients who meet any of the following conditions: a. Patients with anterior wall prolapse of stage III or higher; b. Patients with apical prolapse of stage III or higher;
3. Patients who refuse conservative treatment or have ineffective conservative treatment and request surgical treatment for prolapse;
4. Patients who voluntarily participate in this study, sign the informed consent form, and are able to attend follow-up visits on time;
5. Patients who have received education at the primary school level or above;
6. Patients who are able to visit the hospital for examinations;
7. Patients who are deemed fit to undergo surgery according to preoperative anesthesia assessment.

Exclusion Criteria:

1. Patients who have previously undergone surgery for pelvic organ prolapse (POP);
2. Patients with a history of anti-incontinence surgery or who are planned to undergo mid-urethral sling surgery for anti-incontinence during the current operation;
3. Patients who, after evaluation by the surgeon, have other conditions that affect eligibility for inclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Surgical success rate | From enrollment to the end of surgery at 1 year
  Surgical success is defined as follows:
  1. Points Aa, Ba, Ap, and Bp do not exceed the hymenal margin;
  2. The descent of point C does not exceed one-third of the total vaginal length;
  3. During the follow-up period, the patient does not require pessary treatment or undergo further surgery for pelvic organ prolapse;
  4. Questions 3 of the Pelvic Floor Dysfunction Inventory (PFDI)-20 questionnaire are answered as "none" or "no impact."

SECONDARY OUTCOMES:
Incidence of urinary retention after catheter removal | From enrollment to the end of surgery at 3 days
  A residual urine volume greater than 100 ml as measured by ultrasound is considered urinary retention.
Differences in the severity of overactive bladder (OAB) after surgery | 1 month, 3 months, 6 months and 1 year post-surgery
  It will be assessed by using the Overactive Bladder Symptom Score (OABSS). The score of OABSS ranges from 0 to 15. The higher the score, the more severe the overactive bladder condition is.
Differences in the severity of urinary incontinence after surgery | 1 month, 3 months, 6 months and 1 year post-surgery
  It will be assessed by using the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF). The score of ICIQ-SF ranges from 0 to 21. The higher the score, the more severe the urinary incontinence condition is.
Differences in the severity of pelvic floor dysfunction after surgery | 1 month, 3 months, 6 months and 1 year post-surgery
  It will be assessed using the Pelvic Floor Distress Inventory-20 (PFDI-20).The score of PFDI-20 ranges from 0 to 300. The higher the score, the more severe the pelvic floor dysfunction is.
Differences in quality of life after surgery | 1 month, 3 months, 6 months and 1 year post-surgery
  It will be assessed using the Pelvic Floor Impact Questionnaire (PFIQ).The score of PFIQ ranges from 0 to 300. The higher the score, the poorer the patient's quality of life is.
Differences in patients' satisfaction | 1 month, 3 months, 6 months and 1 year post-surgery
  It will be assessed using the Patient Global Impression of Improvement (PGI-I) questionnaire. The score of PGI-I ranges from 0 to 7. The higher the score, the lower the patient's satisfaction is.
Postoperative Pain | 1 month, 3 months, 6 months and 1 year post-surgery
  It will be assessed using the Wong-Baker Faces Pain Rating Scale (FPS-R). The score of FPS-R ranges from 0 to 10. The higher the score, the more severe the pain is.

OTHER OUTCOMES:
Mesh-related complications | From enrollment to the end of surgery at 1 year
  The Category-Time-Section (CTS) classification is used to document the location, timing, and type of mesh-related complications.
Duration of surgery | Intraoperative
  We record the duration of surgery (hours) based on the anesthesia record sheet.
Blood loss | From enrollment to the end of surgery at 1 year
  We record the amount of blood loss (ml) based on the anesthesia record sheet.
Change in hemoglobin level | From enrollment to the end of surgery at 1 year
  Record the difference in hemoglobin concentration before and after surgery (in g/L).
Hospital stay duration | From enrollment to the end of surgery at 1 year
  The number of days from admission to discharge for the patient (days).
Number of patients with surgical complications | From enrollment to the end of surgery at 1 year
  If patients experience discomfort during the perioperative period or after surgery, they will be advised to seek medical attention promptly to assess for complications. The severity of complications is evaluated using the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes